CLINICAL TRIAL: NCT02657343
Title: An Open-Label, Phase Ib/II Clinical Trial Of Cdk 4/6 Inhibitor, Ribociclib (Lee011), In Combination With Trastuzumab Or T-Dm1 For Advanced/Metastatic Her2-Positive Breast Cancer.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, Sara Tolaney MD, MPH, Dana-Farber Cancer Institute
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15-530; CLEE011XUS20T (Other: Novartis)
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Results first posted 2022-06-03 (Actual); Last update posted 2022-08-01 (Actual); Status verified 2022-07

CONDITIONS: Breast Cancer
Keywords: Breast Cancer With Positive HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — ribociclib; Ado-Trastuzumab Emtansine; Trastuzumab; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Cohort A: Ribociclib + T-DM1 [3+3 Design] (Experimental): * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of Period 1: 300 mg (n = 3), Period 2: 400 mg (n = 3), Period 3: 500 mg (n = 3), and Period 4: 600 mg (n = 3). Maximum dose-escalation of Ribociclib will be up to 600 mg. Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
  Interventions: Drug: Ribociclib; Drug: T-DM1
- Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] (Experimental): * Ribociclib will be given orally once day (400 mg per day on a continuous schedule) for a 21-day cycle of treatment.
  * Trastuzumab will be given as IV infusions over 6 mg/kg every 3 weeks.
  Interventions: Drug: Ribociclib; Drug: Trastuzumab
- Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study] (Experimental): * Ribociclib will be given orally once a day continuously for a 28-day cycle of treatment (except at Dose Level -1, when Ribociclib is given Days 1-21 of a 28 day cycle).
  * Trastuzumab will be given as IV infusions over a pre-determined period of time and dose. Fulvestrant will be dosed approximately every 28 days as per standard of care.
  Interventions: Drug: Ribociclib; Drug: Trastuzumab; Drug: Fulvestrant

INTERVENTIONS:
Drug: Ribociclib
  Other Names: LEE-011
Drug: T-DM1
  Other Names: Kadcyla
  Arms: Cohort A: Ribociclib + T-DM1 [3+3 Design]
Drug: Trastuzumab
  Other Names: Herceptin
  Arms: Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study]; Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study]
Drug: Fulvestrant
  Other Names: Faslodex
  Arms: Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study]

SUMMARY:
Participants that have breast cancer that has spread to other parts of the body, is positive for a protein called HER2, and has not responded to standard treatment. This research study is a way of gaining new knowledge about the combination of Ribociclib with other drugs as a possible treatment for this diagnosis.

DETAILED DESCRIPTION:
This research study is a Phase Ib/II clinical trial, which tests the safety of an investigational intervention and also tries to define the appropriate dose of the investigational intervention to use for further studies.

Ribociclib is a drug that is designed to block certain proteins called Cyclin-Dependent Kinases (CDKs) that are required for cells to divide. These proteins may also control the ability of certain cancers to grow.

In this research study, there will be 3 separate cohorts that are looking for the safe and tolerated dose of ribociclib that can be given in combination with other HER2 directed therapy. One cohort will be looking at the safety of ribociclib in combination with trastuzumab emtansine (T-DM1). T-DM1 is a standard treatment for patients with HER2-positive breast cancer. One Cohort will be looking at the safety of ribociclib in combination with trastuzumab (Herceptin), which is a standard treatment for patients with HER2-positive breast cancer. The last cohort will be looking at the safety of ribociclib in combination with trastuzumab (Herceptin) and fulvestrant (Faslodex) for ER-positive and HER2-positive breast cancer. These are both standard treatments for this type of breast cancer.

The FDA (the U.S. Food and Drug Administration) has not approved Ribociclib as a treatment for any disease.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically confirmed invasive breast cancer, with locally advanced or metastatic disease. Patients without pathologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* The primary tumor, and/or metastasis must have been tested for ER, PR and HER 2, and be HER2 positive as defined by the 2013 ASCO-CAP guidelines.
* Measureable disease by RECIST 1.1 (at least one lesion that can be accurately measured in at least one dimension > 20mm with conventional imaging techniques or > 10mm with spiral CT or MRI) or evaluable disease. Bone lesions (blastic, lytic, or mixed) in the absence of measurable disease as defined above are also acceptable.
* Prior treatment
* Cohort A:

  * Prior treatment with at least one regimen containing Trastuzumab and taxane.
  * No prior treatment with T-DM1 that was discontinued due to disease progression or toxicity.
  * No more than 4 prior lines of therapy in the metastatic setting.
* Cohort B:

  * Must have received prior Trastuzumab, pertuzumab, and T-DM1 in neo-adjuvant, adjuvant, or metastatic setting.
  * No limit on prior lines of therapies.
* Cohort C:

  * Must have received prior Trastuzumab, pertuzumab, and T-DM1 in neo=adjuvant, adjuvant, or metastatic setting.
  * Maximum of 5 prior lines of therapy for metastatic disease.
  * Prior treatment with fulvestrant is permitted.
* Age ≥ 18 years.
* ECOG performance status 0-2 (see Appendix A)
* Participants must have adequate organ and bone marrow function as defined below:

  * Absolute neutrophil count ≥1.5 x 109/L
  * Platelets ≥100 x 109/L
  * Hemoglobin ≥ 9 g/dL
  * Total bilirubin < 1.5xULN; or total bilirubin ≤3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome.
  * Serum creatinine ≤ 1.5 mg/dL or calculated GFR ≥ 50mL/min
  * ALT/AST <2.5x ULN; if liver metastases, ALT/AST ≤5.0x ULN
  * INR ≤ 1.5
  * Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
* Biopsies:

  * Cohorts B and C: all patients with disease that is deemed by the treating investigator as safely accessible to biopsy are required to undergo research biopsies as outlined in this protocol.
  * Cohort A: Such biopsies are optional.
* A negative serum pregnancy test ≤ 72 hours before starting study treatment for premenopausal women and for women < 1 year after the onset of menopause.
* Ability to understand and the willingness to sign a written informed consent document.
* Participants must be able to swallow Ribociclib capsules.
* Patients must have at screening a standard 12-lead ECG with mean values that meet the following parameters:

  * QtcF interval at screening < 450msec (using Friderica's correction)
  * Resting heart rate of 50-90bpm

Exclusion Criteria:

* Participants who have had chemotherapy within 14 days prior registration or those who have not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade ≤1 (Exception to this criterion: patients with any grade of alopecia are allowed to enter the study). There is no washout period required for Trastuzumab.
* Participants who have received radiotherapy ≤ 2 weeks prior to starting study drug, and who have not recovered to grade 1 or better from related side effects of such therapy (except alopecia and neuropathy) and/or in whom ≥ 25% of the bone marrow was irradiated.
* Participants who have previously received a CDK 4/6 inhibitor.
* Participants with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

  * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
  * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to ribociclib, T-DM1 (Cohort A) and/or Trastuzumab (Cohort B).
* In general, the use of any concomitant medication deemed necessary for the care of the patient is permitted in this study, except as specifically prohibited below. Combination administration of study drugs could result in drug-drug interactions (DDI) that could potentially lead to reduced activity or enhanced toxicity of the concomitant medication and/or Ribociclib.
* Patient is currently receiving any of the following medications and cannot discontinue use within 7 days prior to starting study drug (see (Tables 1 and 2, Appendix B for details):

  * Known strong inducers or inhibitors of CYP3A4/5, including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
  * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5
  * Herbal preparations/medications, dietary supplements.
* The list provided here (and in Tables 1 and 2, Appendix B) is not comprehensive and is only meant to be used as a guide. The list is based on the Oncology Clinical Pharmacology Drug-Drug Interaction Database (release date: 29 Oct 2012), which was compiled from the Indiana University School of Medicine's P450 Drug Interaction Table.
* http://medicine.iupui.edu/clinpharm/ddis/main-table/) and supplemented with the FDA Draft Guidance for Industry, Drug Interaction Studies - Study Design, Data Analysis, and Implications for Dosing and Labeling (February 2012) (http://www.fda.gov/downloads/drugs/guidancecomplianceregulatoryinformation/guidances/ucm292362.pdf), and the University of Washington's Drug Interaction Database (http://www.druginteractioninfo.org/). For current lists of medications that may cause QT prolongation and/or torsades de pointes (TdP), refer to the CredibleMeds® website (https://crediblemeds.org/).
* Participants who have any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical trial or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections, etc.).
* Participants who have had major surgery within 2 weeks prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
* Participants who have clinically significant, uncontrolled heart disease and/or cardiac repolarization abnormalities including any of the following:

  * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 6 months prior to screening
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Clinically significant cardiac arrhythmias (e.g. ventricular tachycardia), complete left bundle branch block, high-grade AV block (e.g. bifascicular block, Mobitz type II and third-degree AV block
  * Documented cardiomyopathy
  * Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO) at screening
  * Long QT syndrome or family history of idiopathic sudden death or congenital long QT syndrome, or any of the following

    * Risk factors for Torsades de Pointe (TdP) including uncorrected hypokalemia or hypomagnesemia, history of cardiac failure, or history of clinically significant/symptomatic bradycardia.
    * Inability to determine the QT interval on screening (QTcF, using Fridericia's correction)
  * Systolic blood pressure (SBP)>160 mmHg or <90 mmHg at screening
* Known history of HIV-positivity.
* Active Hepatitis B and/or Hepatitis C Infection
* Known impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., uncontrolled ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection).
* Concurrent malignancy or a malignancy within 3 years prior to starting study drug, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer. Participants with malignancies less than 3 years prior to registration may be considered eligible after discussion with the principle investigator.
* Participants who are currently receiving or have received systemic corticosteroids ≤2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment. The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular).
* Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
* Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer.
* Patient with a Child-Pugh score B or C.
* Participants who have a history of non-compliance to medical therapies.
* Pregnant women are excluded from this study because Ribociclib has the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Ribociclib, breastfeeding should be discontinued if the mother is treated with Ribociclib. These risks also apply to Trasutuzumab used in this study. Pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a postitive hCG laboratory test (>5 mIU/mL).
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Highly effective contraception methods include:

  * Total abstinence when this is in line with the preferred and usual lifestyle of the patient.
  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient
  * Combination of the two following

    * Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    * Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository.
* Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males unless they use a condom during intercourse while taking the drug and for 4 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-03-09 (Actual); Primary Completion 2020-08-27 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD MPH, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Massacusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goel S, Pernas S, Tan-Wasielewski Z, Barry WT, Bardia A, Rees R, Andrews C, Tahara RK, Trippa L, Mayer EL, Winer EP, Spring LM, Tolaney SM. Ribociclib Plus Trastuzumab in Advanced HER2-Positive Breast Cancer: Results of a Phase 1b/2 Trial. Clin Breast Cancer. 2019 Dec;19(6):399-404. doi: 10.1016/j.clbc.2019.05.010. Epub 2019 May 30. PMID 31235441

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 300 mg (n = 3) Maximum dose-escalation of Ribociclib will be up to 600 mg. Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 400 mg (n = 3) Maximum dose-escalation of Ribociclib will be up to 600 mg. Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose: 500 mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 500 mg (n = 3) Maximum dose-escalation of Ribociclib will be up to 600 mg. Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose: 600mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 600 mg (n = 3) Maximum dose-escalation of Ribociclib will be up to 600 mg. Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
Period: Overall Study
Arm/Group | Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg] | Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg] | Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose: 500 mg] | Cohort A: Ribociclib + T-DM1Cohort A: Ribociclib + T-DM1 [Dose: 600mg] | Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] | Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study]
Started | 3 | 3 | 3 | 3 | 13 | 0
Completed | 2 | 1 | 3 | 3 | 12 | 0
Not Completed | 1 | 2 | 0 | 0 | 1 | 0
Not completed — Death | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Patient went to hospice | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: never enrolled to cohort C
Groups:
- Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 300 mg (n = 3) Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 400 mg (n = 3) Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1 [Dose 3: 500mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 500 mg (n = 3) Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Cohort A: Ribociclib + T-DM1 [Dose 4: 600mg]: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 600 mg (n = 3) Dose-escalation will stop if DLT exceed limit.
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
- Total: Total of all reporting groups
Arm/Group | Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg] | Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg] | Cohort A: Ribociclib + T-DM1 [Dose 3: 500mg] | Cohort A: Ribociclib + T-DM1 [Dose 4: 600mg] | Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] | Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study] | Total
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 12 | 0 | 24
Age, Continuous [Median (Full Range); unit: years] | 52 [42 to 59] | 55 [38 to 71] | 52 [37 to 64] | 47 [38 to 62] | 51 [42 to 72] |  | 52 [37 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 3 | 3 | 12 |  | 24
  Male | 0 | 0 | 0 | 0 | 0 |  | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 2 | 2 | 2 | 1 | 12 |  | 19
  Other | 1 | 1 | 1 | 2 | 0 |  | 5
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 3 | 3 | 12 |  | 24

OUTCOME MEASURES:

1. Primary Outcome: Cohort A: Recommended Phase2 Dose (RP2D)
Description: Standard 3+3 phase-I design will be utilized in this trial. Briefly, a minimum of 3 evaluable patients will be entered at first dose level (=300 mg ribociclib) and T-DM1 (3.6 mg/kg IV). If 1 out of the first 3 patients enrolled experiences a dose-limiting toxicity (DLT), 3 additional patients will be enrolled to that dose level. If no more than 1 patient in 6 experiences a DLT, dose escalation of ribociclib will continue to next dose-level. If 2 or more patients at any given dose level experience a DLT, dose escalation will stop and the Recommended Phase2 Dose (RP2D) will be defined. Maximum dose-escalation of Ribociclib (LEE011) will be up to 600 mg.
Time Frame: Disease was evaluated at baseline and each cycle on treatment and the end of treatment. Toxicity was evaluated each cycle on treatment, end of treatment and 30 days follow-up. Median treatment duration was 10.9 months with range 2.5 - 19.3 months.
Measure: Number; unit: mg
Groups:
- Cohort A: Ribociclib + T-DM1: * Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 300 mg (n = 3), 400 mg (n = 3), 500 mg (n = 3), and 600 mg (n = 3).
  * T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 12
mg | 400

2. Primary Outcome: Cohort B: Clinical Benefit Rate (CBR)
Description: CBR is defined as the proportion of patients with a complete response (CR) or partial response (PR), or with stable disease (SD) at week 24 by RECIST 1.1 criteria. CBR will be reported with 90% confidence interval, adjusting for two-stage design using the method from Atkinson and Brown.
Time Frame: at week 12
Measure: Count of Participants; unit: Participants
Groups:
- Cohort B: Ribociclib + Trastuzumab: Ribociclib will be given orally once day continuously for a 21-day cycle of treatment (except at Dose Level -2, when Ribociclib is given Days 1-14 of a 21 day cycle). Trastuzumab will be given as IV infusions over a pre-determined period of time and dose.
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 12
Participants
  CR | 0
  PR | 0
  SD | 3
  Progressive disease | 9

3. Primary Outcome: Cohort C: Clinical Benefit Rate (CBR)
Description: as for outcome 2
Time Frame: at week 12
Population: no patients enrolled
Groups:
- Cohort C: Ribociclib + Trastuzumab + Fulvestrant: * Ribociclib will be given orally once a day continuously for a 28-day cycle of treatment (except at Dose Level -1, when Ribociclib is given Days 1-21 of a 28 day cycle).
  * Trastuzumab will be given as IV infusions over a pre-determined period of time and dose. Fulvestrant will be dosed approximately every 28 days as per standard of care.
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

4. Secondary Outcome: Cohort A: Incidence of Grade 3 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv4 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. median follow-up is 12.4 months
Measure: Number; unit: number of incidences
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 12
number of incidences
  neutropenia | 4
  leukopenia | 4
  anemia | 3
  lymphopenia | 2
  thrombocytopenia | 2
  febrile neutropenia | 1

5. Secondary Outcome: Cohort A: PK Profile of Ribociclib in Combination With T-DM1.
Description: pharmacokinetics (PK) tudies demonstrated dose-related inhibition of Rb phosphorylation in tumors, with continuous dosing over at least 3-5 days being required to achieve optimal target inhibition.
Time Frame: PK blood collection is scheduled at 0 (pre-dose), 0.5, 1, 2, 4, 6, 8, 24 hours following dosing of ribociclib.
Population: 0 patient data collected because study plan changed
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 0

6. Secondary Outcome: Cohort A: Objective Response Rate (ORR)
Description: Objective response rate(ORR) was defined as the portion of patients with complete response or partial response by RECIST 1.1 criteria.
  Complete Response (CR): Disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm. Partial Response (PR): At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Disease was evaluated radiologically at baseline and each cycle on treatment; Treatment continued until disease progression or unacceptable toxicity. Median treatment duration was 10.9 months with range 2.5 - 19.3 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 12
percentage of participants | 16.7 [3 to 44]

7. Secondary Outcome: Cohort A: Median Progression-Free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Disease was evaluated radiologically every cycles on treatment and in long-term follow-up every 12 weeks. Median follow-up in this study cohort was 12.4 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 12
Months | 10.4 [2.7 to 19.3]

8. Secondary Outcome: Cohort A: Frequency of Biomarkers
Description: Optional tumor samples (if safely accessible and feasible) will be taken pre- and post-treatment in order to assess dose-dependent target modulation.
Time Frame: taken at any time in Cycle 2 Day 10-18.
Population: biopsy data not collected because study plan changed
Groups:
- Cohort A: Ribociclib + T-DM1: Ribociclib will be given orally once day (day 5-18) at a pre-determine dose for two weeks of a 21 day cycle. During dose escalation, patients received doses of ribociclib of 300 mg (n = 3), 400 mg (n = 3), 500 mg (n = 3), and 600 mg (n = 3).
  T-DM1 will be given as IV infusions on Day 1 of a 3 week cycle at a pre-determined dose over pre-determined period of time.
Arm/Group | Cohort A: Ribociclib + T-DM1
Number analyzed (Participants) | 0

9. Secondary Outcome: Cohort B: Objective Response Rate (ORR)
Description: as for outcome 6
Time Frame: Disease was evaluated radiologically at baseline and each cycle on treatment; Treatment continued until disease progression or unacceptable toxicity. Median treatment duration was 1.3 months with range 0.6 - 12.6 months.
Measure: Number; unit: rate
Groups:
- Cohort B: Ribociclib + Trastuzumab: * Ribociclib will be given orally once day (400 mg per day on a continuous schedule) for a 21-day cycle of treatment (except at Dose Level -2, when Ribociclib is given Days 1-14 of a 21 day cycle).
  * Trastuzumab will be given as IV infusions over 6 mg/kg every 3 weeks.
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 12
rate | 0

10. Secondary Outcome: Cohort B: Median Progression-Free Survival (PFS)
Description: as for outcome 7
Time Frame: Disease was evaluated radiologically every cycles on treatment and in long-term follow-up every 12 weeks. Median follow-up in this study cohort was 5 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 12
Months | 1.33 [0.92 to 2.57]

11. Secondary Outcome: Cohort B: Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Participants were followed long-term for survival every 12 weeks from the end of treatment until death or lost to follow-up. Median follow-up in this study cohort was 5 months.
Measure: Number (95% Confidence Interval); unit: Months
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 12
Months | 7.9 [3.4 to NA] — based on Kaplan-Meier method limitation, the upper interval cannot be reached

12. Secondary Outcome: Cohort B: Incidence of Grade 3 Treatment-Related Toxicity
Description: as for outcome 4
Time Frame: as for outcome 4
Measure: Number; unit: number of incidences
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 12
number of incidences
  neutropenia | 2
  fatigue | 1
  pain | 1

13. Secondary Outcome: Cohort B: Frequencies Of Biomarkers
Description: as for outcome 8
Time Frame: taken at any time in Cycle 2 Day 10-18.
Population: biopsy will not be done because the study plan changed
Arm/Group | Cohort B: Ribociclib + Trastuzumab
Number analyzed (Participants) | 0

14. Secondary Outcome: Cohort C: Objective Response Rate (ORR)
Description: as for outcome 6
Time Frame: Disease was evaluated radiologically at baseline and each cycle on treatment; Treatment continued until disease progression or unacceptable toxicity. Treatment duration is 0 days since cohort C never enrolled.
Population: data not collected because no patient enrolled
Groups:
- Cohort C: Ribociclib + Trastuzumab + Fulvestrant: Ribociclib will be given orally once a day continuously for a 28-day cycle of treatment (except at Dose Level -1, when Ribociclib is given Days 1-21 of a 28 day cycle). Trastuzumab will be given as IV infusions over a pre-determined period of time and dose. Fulvestrant will be dosed approximately every 28 days as per standard of care.
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

15. Secondary Outcome: Cohort C: Median Progression-Free Survival (PFS)
Description: as for outcome 7
Time Frame: Disease was evaluated radiologically every cycles on treatment and in long-term follow-up every 12 weeks. Reality follow-up is 0 days since cohort C never enrolled.
Population: data not collected because no patients enrolled
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

16. Secondary Outcome: Cohort C: Overall Survival (OS)
Description: as for outcome 11
Time Frame: Participants were followed long-term for survival every 12 weeks from the end of treatment until death or lost to follow-up. 0 days in reality since cohort C never enrolled.
Population: data not collected because no patients enrolled
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

17. Secondary Outcome: Cohort C: Incidence of Grade 3 Treatment-Related Toxicity
Description: as for outcome 4
Time Frame: Assessed each cycle throughout treatment from time of first dose and up to day 30 post-treatment. 0 days in reality since cohort C never enrolled.
Population: data not collected because no patients enrolled
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

18. Secondary Outcome: Cohort C: Frequency of Potential Biomarkers
Description: as for outcome 8
Time Frame: taken at any time in Cycle 2 Day 10-18.
Population: no patients enrolled
Arm/Group | Cohort C: Ribociclib + Trastuzumab + Fulvestrant
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: AE data collected every cycle from the time of the first dose of study treatment, through the study of treatment until 30 days after removal from study or death, whichever occurs first. Cohort A AEs were observed up to 24 weeks, Cohort B AEs were observed up tp 1 cycle (3 weeks).
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg] | Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg] | Cohort A: Ribociclib + T-DM1 [Dose 3: 500mg] | Cohort A: Ribociclib + T-DM1 [Dose 4: 600mg] | Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] | Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study]
All-Cause Mortality (participants affected / at risk) | 0/3 | 2/3 | 0/3 | 0/3 | 0/12 | 0/0
Serious Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 10/12 | 0/0
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 3/3 | 3/3 | 12/12 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 3: 500mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 4: 600mg] (N=3) | Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] (N=12) | Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study] (N=0)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 3 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 1 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 0 | 1 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 1 | 2 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 2 | 2 | 5 | 0
Platelet count decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 0
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 1 | 0
White blood cell decreased (Investigations) | 1 | 1 | 1 | 2 | 4 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A: Ribociclib + T-DM1 [Dose 1: 300mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 2: 400mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 3: 500mg] (N=3) | Cohort A: Ribociclib + T-DM1 [Dose 4: 600mg] (N=3) | Cohort B: Ribociclib + Trastuzumab [Phase 1b/2 Study] (N=12) | Cohort C: Ribociclib + Trastuzumab + Fulvestrant [Phase 1b/2 Study] (N=0)
Activated partial thromboplastin time prolonged (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 1 | 1 | 1 | 1 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 3 | 3 | 2 | 2 | 10 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 1 | 2 | 2 | 0 | 0
Blood bilirubin increased (Investigations) | 2 | 2 | 0 | 0 | 0 | 0
Blurred vision (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 1 | 1 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 1 | 1 | 1 | 0 | 0
Chills (General disorders) | 1 | 1 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 2 | 0 | 0
Cystitis noninfective (Renal and urinary disorders) | 2 | 2 | 0 | 0 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 5 | 0
Dry eye (Eye disorders) | 1 | 1 | 0 | 0 | 2 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 2 | 0
Duodenal hemorrhage (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Edema face (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Electrocardiogram QT corrected interval prolonged (Investigations) | 2 | 2 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 1 | 1 | 0 | 0
Esophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 1 | 1 | 1 | 1 | 0 | 0
Fever (General disorders) | 2 | 2 | 0 | 0 | 0 | 0
Flu like symptoms (General disorders) | 0 | 0 | 1 | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypokalemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0 | 0
Hypomagnesemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0 | 0 | 0
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 2 | 2 | 1 | 1 | 0 | 0
Infections and infestations - Other, specify (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 1 | 0 | 0
Investigations - Other, specify (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Lung infection (Infections and infestations) | 2 | 2 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 1 | 1 | 1 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 2 | 1 | 1 | 5 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 1 | 0 | 0
Nervous system disorders - Other, specify (Nervous system disorders) | 0 | 0 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 3 | 3 | 0 | 0
Oral hemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain (General disorders) | 0 | 0 | 2 | 2 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Platelet count decreased (Investigations) | 3 | 3 | 3 | 3 | 0 | 0
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Scalp pain (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0
Skin infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 2 | 2 | 0 | 0 | 0 | 0
Watering eyes (Eye disorders) | 0 | 0 | 1 | 1 | 1 | 0
Weight gain (Investigations) | 1 | 1 | 0 | 0 | 0 | 0
Weight loss (Investigations) | 2 | 2 | 0 | 0 | 0 | 0
White blood cell decreased (Investigations) | 3 | 3 | 2 | 2 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02657343/Prot_SAP_000.pdf